CLINICAL TRIAL: NCT04565561
Title: Neovas Versus DCB for Coronary de Novo Lesions in Patients With STEMI: a Prospective Observational Clinical Trial
Brief Title: Bioabsorbable Scaffold vs Drug-coated Balloon for Coronary de Novo Lesions in STEMI: Prospective Observational Trial
Acronym: NeovasvsDCB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY-LL-2020099-02
Record Dates: First submitted 2020-09-23; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Diseases
Keywords: Neovas BRS; DCB; DES; STEMI
MeSH Terms: conditions — Cardiovascular Diseases; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neovas BRS group: Neovas BRS group, n=20
  Interventions: Device: Neovas BRS or DCB
- DCB group: DCB group, n=20
  Interventions: Device: Neovas BRS or DCB

INTERVENTIONS:
Device: Neovas BRS or DCB — All STEMI patients were predilated (including predilated balloon or cutting balloon) before randomization. Thrombus aspiration was determined by the surgeon according to the specific situation.
  Sufficient predilation criteria: the following two conditions must be met: A. residual stenosis < 30%; B. no flow limiting dissection or TIMI grade 2-3.
  Other Names: DES

SUMMARY:
a prospective, single center, observational clinical trail. Aim to to compare the efficacy and safety of the Bioabsorbable scaffold (BRS) Neovas BRS and Drug-coating balloon (DCB) in the treatment of STEMI patients with coronary artery disease and to further evaluate the safety and effectiveness of the two new interventional methods in STEMI intervention, so as to better guide clinical practice.

DETAILED DESCRIPTION:
1. To study the advantages and disadvantages of Neovas BRS and DCB in interventional treatment of de novo lesions in STEMI patients, in order to better guide the clinical.
2. To explore the safety of Neovas BRS in interventional treatment of ide novo lesions in STEMI patients.
3. To explore the safety of DCB in interventional treatment of de novo lesions in STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

1) Age > 18 years old (2) STEMI patients suitable for PPCI operation. Chest pain for more than 20 minutes; At least 2 leads ST-T segment elevation > 1 mm, or new LBBB, or myocardial infarction confirmed by echocardiography; It is expected that the reperfusion treatment can be successfully implemented within 12 hours after the occurrence of acute myocardial infarction.

(3) Target vessels are suitable for PPCI and Single vessel disease (non culprit vessel stenosis < 50%). It is a primary coronary lesion; Reference vessel diameter > 2.5mm and < 4mm, lesion length < 20mm; There is no obvious calcification at the lesion site; After thrombus aspiration or pre dilation balloon pretreatment, the residual stenosis < 30% has no blood flow restrictive dissection.

(4) Patients refused to accept drug-eluting stent implantation, voluntarily participated and signed informed consent, accepted and was willing to cooperate with follow-up, and was willing to cooperate with standard secondary prevention and treatment of coronary heart disease.

Exclusion Criteria:

The age is less than 18 years old; Previous history of myocardial infarction or post coronary stent operation; Left main disease; It is known that it is contraindications or resistance to the following drugs: bevaludine, low molecular heparin, common heparin, aspirin, clopidogrel / tegrelol; Participate in other clinical studies and interfere with the study; It is uncertain whether there is any neurological injury: for example, after resuscitation; It needs tracheal intubation / artificial ventilation; There was cardiogenic shock before grouping; It is known that there are intracranial diseases: occupying position, aneurysm, arteriovenous malformation, hemorrhagic cerebrovascular accident, ischemic cerebrovascular accident; Internal bleeding such as gastrointestinal bleeding before selection; It is planned to perform major surgical treatment within 6 weeks; Serious infectious disease, malignant tumor disease, serious blood disease and autoimmune disease; in recent March, there has been a history of large-dose use of immunosuppressant; Non coronary vasculitis and thrombotic diseases (vasculitis, aortic dissection, abdominal aneurysm); Serious mental illness patients; The life expectancy is less than 1 year; No consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients undergoing PPCI
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
late lumen loss (LLL) | 1-year
  The primary endpoint in-segment is late lumen loss (LLL) with follow-up of 1 year.

SECONDARY OUTCOMES:
target lesion revascularization (TLR) | 1-year
  The secondary endpoint is target lesion revascularization (TLR) with follow-up of 1 year.
cardiac death | 1-year
  The secondary endpoint is cardiac death with follow-up of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: yaowang lin, master, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No